CLINICAL TRIAL: NCT02041234
Title: Roux-en-Y Gastric Bypass for BMI 27-32 Type 2 Diabetes vs Best Medical Treatment
Brief Title: Roux-en-Y Gastric Bypass for BMI 27-32 Type 2 Diabetes Versus Best Medical Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Anton Cheng, Dr Anton Cheng, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bariatric Surgery RCT
Record Dates: First submitted 2014-01-10; First posted 2014-01-22 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Type II Diabetes in Subjects BMI 27 to 32
Keywords: Diabetes; surgical treatment; medical treatment
MeSH Terms: conditions — Diabetes Mellitus | interventions — Gastric Bypass; Liraglutide; Orlistat; Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; Canagliflozin; Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y Gastric Bypass (RYGB) (Active Comparator): Roux-en-Y Gastric Bypass (RYGB) as per standard surgical protocol, with a 30 cc gastric pouch, 50 cm biliopancreatic limb and 100cm gastrointestinal limb.
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB)
- Best Medical Treatment (Active Comparator): Anti-diabetic medications provided (Mono- or Combination- therapy):
  Incretin analogues: Liraglutide up to 3 mg daily Or DPP-4 Inhibitors: Sitagliptin up to 100 mg daily, Linagliptin up to 5mg daily Xenical: Up to 120 mg tds SGLT2 inhibitors: Empagliflozin up to 25mg daily, Canagliflozin up to 300mg daily Participants will also take lipids & BP medications according to standard of care.
  Interventions: Drug: Incretin analogues; Drug: Xenical; Drug: SGLT2 inhibitors; Drug: DPP-4 Inhibitors

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGB) — Roux-en-Y Gastric Bypass (RYGB) as per standard surgical protocol, with a 30 cc gastric pouch, 50 cm biliopancreatic limb and 100cm gastrointestinal limb.
  Arms: Roux-en-Y Gastric Bypass (RYGB)
Drug: Incretin analogues — Incretin analogues: Liraglutide up to 1.8 mg daily
  Other Names: Liraglutide
  Arms: Best Medical Treatment
Drug: Xenical — Xenical: Up to 120 mg tds
  Other Names: Orlistat
  Arms: Best Medical Treatment
Drug: SGLT2 inhibitors — SGLT2 inhibitors: Empagliflozin up to 25mg daily, Canagliflozin up to 300mg daily
  Other Names: Empagliflozin; Canagliflozin
  Arms: Best Medical Treatment
Drug: DPP-4 Inhibitors — Sitagliptin up to 100 mg daily, Linagliptin up to 5mg daily
  Other Names: Sitagliptin; Linagliptin
  Arms: Best Medical Treatment

SUMMARY:
Investigators aim to show that Roux-en-Y Gastric Bypass (RYGB) is superior to best medical treatment in reaching well-defined treatment end points in Asian subjects of BMI 27-32 with type 2 Diabetes (DM2). Investigators also hope to show that successful RYGB will reduce resource utilization in the near term with similar projected reduction over the medium to long term.

DETAILED DESCRIPTION:
40 subjects with DM2 will be recruited, randomised into two arms. The surgical arm will be subjected to RYGB. The medical arm will be treated maximally utilising the best means available and following internationally available protocol/guidelines. The study population will be subjected to a set of tests which is over and above the standard tests for similar groups of patients undergoing standard care (details below). Some test samples will be bio-banked. Treatment end points and follow up protocol will be the same for each treatment arm. The International Diabetic Federation (IDF) in 2011 recommended that bariatric surgery should be considered an alternative treatment option for those Asian DM2 subjects with BMI of 27 or above. Data for the effectiveness of Bariatric Surgery for those DM subjects with lower BMI is not as well established as those with higher BMI. There is scant good quality data, especially from Asian subjects. As their treatment is totally funded by the research project, subjects on the non surgical treatment arm will benefit from the more intense management of their disease with no restriction due to cost. The surgical arm will also be fully funded by the research project. They will be exposed to the standard risks associated with this type of surgery. Subjects in both arms will have to provide more blood and other samples than usual and has to follow visits protocol as close as possible. RYGB is a major surgical procedure, with significant potential complications; during the process of surgery and afterwards, both short and long term. Procedure related mortality is about 0.3%. Major complications that may require surgical intervention includes: anastomotic leakage about 3-4%, bleeding 3%, infection 3%, venous thrombo-embolism 1%. Some of these complications will require prolong hospitalisation. After surgery, loose stool, dumping syndrome, anastomotic ulcers can occur in less than 3%.Life long dietary supplement will be required. Longer term post surgical complications include intestinal obstruction due to adhesions or internal hernia, about 2%, further surgery may be needed. This risk is lifelong. Nutritional deficiencies, especially if not compliant with regular supplement intake, may occur. Drug allergies can occur; from simple rash to life threatening anaphylactic reaction. Blood taking can cause bruising, pain at the puncture site and sometimes fainting.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of DM2 = or < 10 years
2. Age 21-65
3. BMI 27-32.
4. HBA1c ≥ 8%, on maximum treatment from primary care physician
5. At least one of the following co-morbidities on treatment: hypertension, hyperlipidaemia, micro/macro-proteinuria or ≤class I nephropathy, retinopathy.

Exclusion Criteria:

1. Subjects who had previous Bariatric surgery or extensive upper abdominal surgery
2. Pregnant subjects.
3. Nephropathy requiring dialysis
4. Subjects who are not fit for general anaesthesia.
5. Subjects who are unsuitable for RYGB for whatever reason, medical/surgical/psychological.
6. Subjects who are unwilling or possibly unable to participate in the follow up process.
7. Subjects who are reluctant to be randomised into the two study groups.
8. Subjects who suffers from unstable psychiatric illness
9. Subjects who are active substance abusers
10. Glutamic acid decarboxylase antibody positive.
11. fasting C-peptide < 300 pmol/L

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2020-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving HBA1c of 6% without diabetic medication | at 12 month after randomisation
  The primary endpoint is to compare Roux-en-Y Gastric Bypass (RYGB) vs best medical treatment for Asian subjects of BMI 27-32 with poorly controlled type 2 Diabetes (DM2) in achieving a glycated haemoglobin level of 6% or less at 12 months after randomisation, and beyond till the end of the study period, without diabetic medications; and also systolic Blood Pressure of <130 mm HG, and LDL of <100mg/dl.
Number of subjects achieving systolic BP <130mm hg without antihypertension medication | 12 months post randomisation
  The primary endpoint is to compare Roux-en-Y Gastric Bypass (RYGB) vs best medical treatment for Asian subjects of BMI 27-32 with poorly controlled type 2 Diabetes (DM2) in achieving a glycated haemoglobin level of 6% or less at 12 months after randomisation, and beyond till the end of the study period, without diabetic medications; and also systolic Blood Pressure of <130 mm HG, and LDL of <100mg/dl.
number of subjects achieving LDL level of <100mg/dl without lipid lowering medication | 12 months post randomisation
  The primary endpoint is to compare Roux-en-Y Gastric Bypass (RYGB) vs best medical treatment for Asian subjects of BMI 27-32 with poorly controlled type 2 Diabetes (DM2) in achieving a glycated haemoglobin level of 6% or less at 12 months after randomisation, and beyond till the end of the study period, without diabetic medications; and also systolic Blood Pressure of <130 mm HG, and LDL of <100mg/dl.

SECONDARY OUTCOMES:
fasting plasma glucose | 12 months after Randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
Fasting Insulin | 12 months after radomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
serum c-peptide level | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
serum lipid levels | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
C-reactive protein level | 12 months post randolmisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
change in medications usage | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
changes in gut hormones levels | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
changes in metabolic hormones level | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
health resource utilisation | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
  On medium term follow up, we hope to evaluate the effect of successful DM2 improvement post surgery results in reduced resource utilization in the near term and a similar projected reduction over the long term.
HOMA-IR | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
Blood Pressure measurement | 12 months post randomisation
number of adverse events | 12 months post randomisaiton
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.
Weight loss | 12 months post randomisation
  Secondary end points include levels of fasting plasma glucose, fasting insulin, C-peptide, lipids, C-reactive protein (CRP), the homeostasis model assessment of insulin resistance (HOMA-IR) index, weight loss, blood pressure, adverse events, changes in medications, serum gut hormones and metabolic hormone levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Cheng, MBBS, Principal Investigator — Khoo Teck Puat Hospital; Su Chi Lim, MBBS, PhD, Principal Investigator — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colquitt JL, Picot J, Loveman E, Clegg AJ. Surgery for obesity. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003641. doi: 10.1002/14651858.CD003641.pub3. PMID 19370590
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Dixon JB, Zimmet P, Alberti KG, Rubino F; International Diabetes Federation Taskforce on Epidemiology and Prevention. Bariatric surgery: an IDF statement for obese Type 2 diabetes. Diabet Med. 2011 Jun;28(6):628-42. doi: 10.1111/j.1464-5491.2011.03306.x. PMID 21480973
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Background] Cohen RV, Pinheiro JC, Schiavon CA, Salles JE, Wajchenberg BL, Cummings DE. Effects of gastric bypass surgery in patients with type 2 diabetes and only mild obesity. Diabetes Care. 2012 Jul;35(7):1420-8. doi: 10.2337/dc11-2289. PMID 22723580
- [Derived] Cheng A, Yeoh E, Moh A, Low S, Tan CH, Lam B, Sum CF, Subramaniam T, Lim SC. Roux-en-Y gastric bypass versus best medical treatment for type 2 diabetes mellitus in adults with body mass index between 27 and 32 kg/m2: A 5-year randomized controlled trial. Diabetes Res Clin Pract. 2022 Jun;188:109900. doi: 10.1016/j.diabres.2022.109900. Epub 2022 May 2. PMID 35513159